CLINICAL TRIAL: NCT01986257
Title: Emotion Regulation Group Therapy (ERGT) for Women Engaging in Non-suicidal Self-Injury (NSSI) - an Effectiveness Study
Brief Title: ERGT for Women Engaging in NSSI - an Effectiveness Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Clara Hellner Gumpert, Ph.D., Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DNR 2013/1321-31/3
Record Dates: First submitted 2013-11-04; First posted 2013-11-18 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Borderline Personality Disorder; Non-suicidal Self-injury (NSSI)
MeSH Terms: conditions — Borderline Personality Disorder; Self-Injurious Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Emotion Regulation Group Therapy (ERGT). (Experimental)
  Interventions: Behavioral: Emotion Regulation Group Therapy (ERGT).

INTERVENTIONS:
Behavioral: Emotion Regulation Group Therapy (ERGT).

SUMMARY:
The primary aim is to investigate the effectiveness of Emotion Regulation Group Therapy (ERGT) for women who self-harm in ordinary psychiatric outpatient health care.

ELIGIBILITY:
Inclusion Criteria:

* NSSI a minimum of three times in the last six months
* Meets at least three criteria for Borderline Personality Disorder according to DSM-IV-TR
* Contact with an other individual therapist, psychiatrist, "case manager" or equal

Exclusion Criteria:

* Insertion/withdrawal of psychopharmacological substances within two months prior to the treatment
* Other acute primary axis I diagnosis (e.g. anorexia nervosa) that demand treatment in first hand
* Bipolar disorder I or primary psychosis
* Current substance dependence (the last month)
* Current life circumstances that would hinder the treatment (i.e. ongoing domestic abuse)
* Insufficient Swedish language skills
* Cocurrent treatment with Mentalization based therapy (MBT) or Dialectical behavioral therapy (DBT)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Frequency of non-suicidal self-injury as measured by Deliberate Self-Harm Inventory (DSHI) | Baseline (from inclusion to treatment start), (7 days prior to treatment start), weekly (once a week following treatment start), post-treatment (14 weeks) and six and twelve months follow-up.
  Change from Baseline in deliberate self-harm after 14 weeks and at 6- and 12 months after treatment has ended.

SECONDARY OUTCOMES:
Borderline Symptom List Behavior supplement (BSL-supplement) | Baseline (from inclusion to treatment start), pre-treatment (7 days prior to treatment start), weekly (once a week following treatment start), post-treatment (14 weeks), and six and twelve months follow-up.
  Change from Baseline in self-destructive behaviors after 14 weeks and at 6- and 12 months after treatment has ended.
Difficulties in Emotion Regulation Scale (DERS) | Baseline (from inclusion to treatment start), pre-treatment (7 days prior to treatment start), weekly (once a week following treatment start), post-treatment (14 weeks) and six and twelve months follow-up.
  Change from Baseline in difficulties with emotion regulation after 14 weeks and at 6- and 12 months after treatment has ended.
Diary questionnaire (DQ) | Baseline (from inclusion to treatment start), pre-treatment (7 days prior to treatment start), weekly (once a week following treatment start), post-treatment (14 weeks) and six and twelve months follow-up.
  Change from Baseline in positive and negative affect after 14 weeks and at 6- and 12 months after treatment has ended.
The Borderline Evaluation of Severity over Time (BEST). | Pre-treatment (7 days prior to treatment start), post-treatment (14 weeks) and six and twelve months follow-up.
  Change from Baseline in Borderline severity symptoms after 14 weeks and at 6- and 12 months after treatment has ended.
The Depression Anxiety Stress Scales (DASS) | Pre-treatment (7 days prior to treatment start), post-treatment (14 weeks) and six and twelve months follow-up.
  Change from Baseline in depression and anxiety after 14 weeks and at 6- and 12 months after treatment has ended.
Inventory of Interpersonal Problems - Borderline Personality Disorder (IIP-BPD) | Pre-treatment (7 days prior to treatment start), post-treatment (14 weeks) and six and twelve months follow-up.
  Change from Baseline in interpersonal problems after 14 weeks and at 6- and 12 months after treatment has ended.
Sheehan Disability Scale (SDS) | Pre-treatment (7 days prior to treatment start), post-treatment (14 weeks) and six and twelve months follow-up.
  Change from Baseline in global functioning after 14 weeks and at 6- and 12 months after treatment has ended.
Trimbos and Institute of Technology Cost Questionnaire for Psychiatry (TIC-P) | Baseline, post-treatment (14 weeks) and six and twelve months follow-up.
  Change from Baseline in societal costs after 14 weeks and at 6- and 12 months after treatment has ended.
Euroqol-5D (EQ-5D) | Baseline, post-treatment (14 weeks) and six and twelve months follow-up.
  Change from Baseline in quality of life after 14 weeks and at 6- and 12 months after treatment has ended.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Psychiatry Research Karolinska Institutet and Stockholm County Council, Stockholm, Sweden

REFERENCES:
- [Derived] Sahlin H, Bjureberg J, Gratz KL, Tull MT, Hedman E, Bjarehed J, Jokinen J, Lundh LG, Ljotsson B, Hellner C. Emotion regulation group therapy for deliberate self-harm: a multi-site evaluation in routine care using an uncontrolled open trial design. BMJ Open. 2017 Oct 5;7(10):e016220. doi: 10.1136/bmjopen-2017-016220. PMID 28982814